CLINICAL TRIAL: NCT07127640
Title: Effect of an Aerobic Exercise Session on Cardiovascular and Autonomic Parameters of Adults With Hypertrophic Cardiomyopathy: a Randomized Clinical Trial
Brief Title: Effect of an Aerobic Exercise Session on Cardiovascular and Autonomic Parameters of Adults With Hypertrophic Cardiomyopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UP 6126/24
Record Dates: First submitted 2025-05-30; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cardiomyopathy, Hypertrophic; Physical Exercise; Autonomic Nervous System; Endothelium; Blood Pressure
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): An aerobic exercise session on a recumbent exercise bike with a 5-minute warm-up period, followed by a 40-minute cool-down period and ending with a 5-minute cool-down at decreasing speed.
  Interventions: Other: Exercise
- Control (No Intervention): The control session will consist of the individual remaining seated for 50 minutes in an air-conditioned room.

INTERVENTIONS:
Other: Exercise — An aerobic exercise session on a recumbent exercise bike with a 5-minute warm-up period, followed by a 40-minute cool-down period and ending with a 5-minute cool-down at decreasing speed.
  Arms: Exercise

SUMMARY:
Hypertrophic cardiomyopathy is a genetic heart disease with symptoms that may include dyspnea and fatigue predominantly on exertion, with or without chest pain, palpitations, syncope/presyncope and sudden cardiac death, mostly in young individuals, often without symptoms. Due to the higher cardiovascular risk described for individuals with hypertrophic cardiomyopathy, it is extremely important to create non-pharmacological strategies that can minimize the evolution of cardiovascular risk factors found in this population. The objective of the study will be to evaluate the effect of an aerobic exercise session on the ratio between the low frequency (LF) and high frequency (HF) bands of heart rate variability, endothelial function through flow-mediated dilation and systolic and diastolic blood pressure during the 24-hour period in adult individuals with hypertrophic cardiomyopathy. The study design will be a randomized crossover clinical trial with individuals aged 18 to 59 years, of both sexes, randomized by lottery and divided into two groups: Exercise group and control group without exercise. An exercise stress test will be performed and on a new date the individuals will perform a supervised session of moderate-intensity aerobic exercise on a horizontal stationary bicycle for 50 minutes or will remain seated in an air-conditioned room for the same period of time. Subsequently, the procedures will be crossed. It is expected to find improvements in the parameters of endothelial function, autonomic modulation and 24-hour blood pressure in adult individuals with non-obstructive hypertrophic cardiomyopathy undergoing a session of aerobic physical exercise when compared to a control session without exercise.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of individuals aged between 18 and 59 years with HCM diagnosed via ICFUC medical records.

Exclusion Criteria:

* Individuals with a history of exercise-induced arrhythmias, a history of aborted sudden death, and the presence of an implantable cardioverter defibrillator will be excluded from the sample. Those with LVOT obstruction at rest ≥50 mmHg on medical therapy, recent septal reduction therapy, pregnancy, class IV symptoms in the New York Heart Association (NYHA) functional classification78, hypotensive response to exercise (drop in systolic BP >20 mmHg in relation to the resting value or during exercise) will also be excluded. Concomitantly, those with systolic dysfunction of left ventricular ejection fraction <50%, myocardial infarction, or previous stroke will be excluded. Hypertensive patients, those with orthopedic limitations, or any physical or mental limitation that prevents them from performing physical exercises will also be excluded.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of autonomic system function | From enrollment to the end of treatment at 2 weeks
  Ratio between the low frequency (LF) and high frequency (HF) bands of heart rate variability by electrocardiogram

SECONDARY OUTCOMES:
Assessment of endothelial function | From enrollment to the end of treatment at 2 weeks
  Flow-mediated dilation (FMD) by high-resolution Doppler ultrasound images of the brachial artery.
Blood pressure assessment | From enrollment to the end of treatment at 2 weeks
  Ambulatory Blood Pressure Monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia do Instituto de Cardiologia do Rio Grande do Sul / Fundação Universitária de Cardiologia (IC/FUC)o Grande do Sul / Fundação Universitária de Cardiologia (IC/FUC), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No